CLINICAL TRIAL: NCT02243696
Title: Protego DF4 Post Approval Registry
Status: Terminated | Type: Observational
Why Stopped: On April 15, 2019, BIOTRONIK received FDA approval to transition the ongoing Protego DF4 Post Approval Registry to a new EP PASSION real-world data methodology.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P980023/S057
Record Dates: First submitted 2014-09-11; First posted 2014-09-18 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Implantable Defibrillator User

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry study is to confirm the long-term safety and reliability of the Protego DF4 right ventricular lead.

ELIGIBILITY:
Inclusion Criteria:

* Implanted within the last 30 days or candidate for implantation of a BIOTRONIK ICD or CRT-D DF4 compatible system along with the Protego DF4 lead
* Meets ICD or CRT-D system implant recommendations as defined in guidelines published by relevant professional societies
* Able to understand the nature of the registry and provide informed consent
* Available for follow-up visits on a regular basis at the investigational site for the expected 5 years of follow-up
* Age greater than or equal to 18 years

Exclusion Criteria:

* Enrolled in any investigational cardiac device trial
* Planned cardiac surgical procedures or interventional measures within the next 6 months
* Expected to receive heart transplantation or ventricular assist device within 1 year
* Life expectancy of less than 1 year
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Patients reporting pregnancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigators' general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1694 (Actual)
Dates: Start 2014-09-27 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (68):
  - Gadsden, Alabama
  - Avondale, Arizona
  - Glendale, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Escondido, California
  - Fountain Valley, California
  - Hawthorne, California
  - Los Angeles, California
  - Santa Barbara, California
  - Temecula, California
  - Torrance, California
  - Norwalk, Connecticut
  - Brooksville, Florida
  - Daytona Beach, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Smyrna Beach, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Alton, Illinois
  - Aurora, Illinois
  - Chicago, Illinois
  - Schaumburg, Illinois
  - Fort Wayne, Indiana
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Lafayette, Louisiana
  - Lake Charles, Louisiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Flint, Michigan
  - Lansing, Michigan
  - Rochester Hills, Michigan
  - Wyoming, Michigan
  - Ypsilanti, Michigan
  - St Louis, Missouri
  - Clifton, New Jersey
  - Mineola, New York
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Middletown, Ohio
  - Steubenville, Ohio
  - Philadelphia, Pennsylvania
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Lancaster, South Carolina
  - Mt. Pleasant, South Carolina
  - Rock Hill, South Carolina
  - Corpus Christi, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Kingwood, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Fredericksburg, Virginia
  - Norfolk, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOTRONIK Protego DF4 Lead: Patients with a Protego DF4 lead used in conjunction with any market-released BIOTRONIK ICD or cardiac resynchronization therapy defibrillator device with a DF4 header.
Period: Overall Study
Arm/Group | BIOTRONIK Protego DF4 Lead
Started | 1694
Completed | 0
Not Completed | 1694
Not completed — Death | 282
Not completed — Withdrawal by Subject | 79
Not completed — Lost to Follow-up | 57
Not completed — Subject No Longer has Study System | 42
Not completed — Subject Withdrawn by Investigator | 273
Not completed — Study Terminated for EP PASSION | 961

BASELINE CHARACTERISTICS:
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481
  Male | 1213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 177
  Not Hispanic or Latino | 1326
  Unknown or Not Reported | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 340
  White | 1130
  More than one race | 0
  Unknown or Not Reported | 181
Weight [Mean (Standard Deviation); unit: pounds] — Population: Baseline characteristics are provided when available, subjects without an available baseline characteristic are not included in the number of participants analyzed for that characteristic.
  pounds
    number analyzed (Participants) | 1656
    (all) | 196.3 (51.28)
Height [Mean (Standard Deviation); unit: inches] — Population: Baseline characteristics are provided when available, subjects without an available baseline characteristic are not included in the number of participants analyzed for that characteristic.
  inches
    number analyzed (Participants) | 1653
    (all) | 67.7 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With No Protego DF4 Lead Adverse Event
Description: Evaluate the percentage of subjects without an adverse event related to the Protego DF4 lead or header through 5 years. The endpoint is analyzed as the adverse event free-rate.
Time Frame: Up to 4.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
percentage of participants | 98.7 [98.04 to 99.18]

2. Primary Outcome: Protego DF4 Lead Safety-Individual Adverse Event-Free Rate
Description: Evaluate the individual types of adverse events contributing to primary outcome measure 'Protego DF4 Lead Safety-Overall Adverse Event-Free Rate'.
Time Frame: Up to 4.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
percentage of participants
  Lead oversensing | 0.41 [0.17 to 0.85]
  Lead conductor fracture | 0.30 [0.10 to 0.69]
  Lead dislodgement | 0.18 [0.03 to 0.55]
  Lead impedance our of range, high | 0.12 [0.01 to 0.43]
  Lead impedance out of range, low | 0.12 [0.01 to 0.43]
  Cardiac perforation | 0.06 [0.01 to 0.33]
  Inability to extend helix | 0.06 [0.01 to 0.33]
  Lead failure | 0.06 [0.01 to 0.33]

3. Secondary Outcome: Protego DF4 Lead Pacing Threshold Measurement
Description: Pacing threshold measurements at pulse width of 0.4 or 0.5 ms for the Protego DF4 leads through 5 years of follow-up.
Time Frame: Up to 4.5 years
Population: A threshold measurement for the Protego lead using a pulse width of 0.4 or 0.5 ms was unavailable for one subject. This patient was excluded from the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1693
volts | 0.67 (0.36)

4. Secondary Outcome: Protego DF4 Lead Shock Impedance
Description: Shock impedance measurements for the Protego DF4 leads through 5 years of follow-up.
Time Frame: Up to 4.5 years
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
Ohms | 71.5 (13.4)

5. Secondary Outcome: Percentage of Subjects With no Adverse Events Excluded From Primary Objectives
Description: The overall percentage of patients without adverse events that were excluded from the primary objectives and occurred through 5 years of follow-up. This was evaluated as an adverse event free-rate (AEFR).
Time Frame: Up to 4.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
percentage of participants | 90.73 [89.25 to 92.07]

6. Secondary Outcome: Protego DF4 Lead Sensing
Description: Sensing measurements for the Protego DF4 leads through 5 years of follow-up.
Time Frame: Up to 4.5 years
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
millivolts | 15.70 (5.97)

7. Secondary Outcome: Protego DF4 Lead Pacing Impedance
Description: Pacing impedance measurements for the Protego DF4 leads through 5 years of follow-up.
Time Frame: Up to 4.5 years
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | BIOTRONIK Protego DF4 Lead
Number analyzed (Participants) | 1694
Ohms | 552.3 (121.5)

ADVERSE EVENTS:
Time Frame: Up to 4.5 years
Description: According to the study protocol, sites were required to report all patient deaths and all adverse events that were considered related to the implant procedure, implanted pulse generator, or implanted leads. Adverse events determined to be not related to the implant procedure, implanted pulse generator, or implanted leads were not collected.
  Reported adverse events were defined as a serious or 'other' adverse event according to the clinicaltrials.gov definition.
Arm/Group | BIOTRONIK Protego DF4 Lead
All-Cause Mortality (participants affected / at risk) | 282/1694
Serious Adverse Events (participants affected / at risk) | 145/1694
Other Adverse Events (participants affected / at risk) | 144/1694
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Protego DF4 Lead (N=1694)
Atrial lead conductor fracture (Cardiac disorders) | 2 (2)
Atrial lead dislodgement (Cardiac disorders) | 21 (21)
Atrial lead high pacing threshold (Cardiac disorders) | 1 (1)
Cardiac perforation (Cardiac disorders) | 2 (2)
Inability to defibrillate successfully with the Protego lead (Cardiac disorders) | 1 (1)
LV lead diaphragmatic stimulation (Cardiac disorders) | 5 (5)
LV lead dislodgement (Cardiac disorders) | 6 (7)
LV lead high pacing threshold (Cardiac disorders) | 3 (3)
LV lead impedance out of range, high impedance (Cardiac disorders) | 1 (1)
LV lead intermittent capture / no lead capture (Cardiac disorders) | 2 (2)
Premature battery depletion (Cardiac disorders) | 3 (3)
Pulse generator failure (Cardiac disorders) | 1 (1)
Pulse generator migration (Cardiac disorders) | 1 (1)
RV lead conductor fracture (Cardiac disorders) | 6 (6)
RV lead dislodgement (Cardiac disorders) | 26 (27)
RV lead failure (Cardiac disorders) | 1 (1)
RV lead high pacing threshold (Cardiac disorders) | 5 (5)
RV lead impedance out of range, high impedance (Cardiac disorders) | 5 (5)
RV lead impedance out of range, low impedance (Cardiac disorders) | 4 (4)
RV lead intermittent capture / no lead capture (Cardiac disorders) | 2 (2)
RV lead oversensing not due to external noise (Cardiac disorders) | 9 (9)
RV lead undersensing or loss of sensing (Cardiac disorders) | 3 (3)
Pulmonary embolism (General disorders) | 1 (1)
Twiddler's syndrome (General disorders) | 2 (2)
Primary infection (Infections and infestations) | 21 (21)
Secondary infection (Infections and infestations) | 7 (7)
Skin erosion (Skin and subcutaneous tissue disorders) | 2 (2)
Cardiac perforation with or without tamponade (Surgical and medical procedures) | 2 (2)
Coronary sinus dissection (Surgical and medical procedures) | 2 (2)
Hematoma (Surgical and medical procedures) | 9 (9)
Loose set-screw (Surgical and medical procedures) | 2 (2)
Pneumothorax (Surgical and medical procedures) | 3 (3)
Pocket pain (Surgical and medical procedures) | 1 (1)
Pulmonary embolism (Surgical and medical procedures) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Protego DF4 Lead (N=1694)
Atrial lead dislodgement (Cardiac disorders) | 5 (5)
Atrial lead high pacing threshold (Cardiac disorders) | 13 (13)
Atrial lead impedance out of range, high impedance (Cardiac disorders) | 3 (3)
Atrial lead impedance out of range, low impedance (Cardiac disorders) | 1 (1)
Atrial lead intermittent capture / no lead capture (Cardiac disorders) | 1 (1)
Bent connector pin noted during implant procedure (Cardiac disorders) | 2 (2)
Inability to extend helix during implant procedure (Cardiac disorders) | 3 (3)
Inability to successfully implant Protego lead (Cardiac disorders) | 1 (1)
LV lead diaphragmatic stimulation (Cardiac disorders) | 31 (38)
LV lead dislodgement (Cardiac disorders) | 1 (1)
LV lead high pacing threshold (Cardiac disorders) | 59 (67)
LV lead impedance out of range, high impedance (Cardiac disorders) | 1 (1)
LV lead intermittent capture / no lead capture (Cardiac disorders) | 5 (6)
LV lead oversensing not due to external noise (Cardiac disorders) | 1 (1)
Pulse generator back-up mode initiated (Cardiac disorders) | 5 (5)
RV lead diaphragmatic stimulation (Cardiac disorders) | 1 (1)
RV lead high pacing threshold (Cardiac disorders) | 10 (10)
RV lead impedance out of range, high impedance (Cardiac disorders) | 1 (1)
RV lead impedance out of range, low impedance (Cardiac disorders) | 1 (1)
RV lead intermittent capture / no lead capture (Cardiac disorders) | 1 (1)
RV lead oversensing not due to external noise (Cardiac disorders) | 3 (3)
RV lead undersensing or loss of sensing (Cardiac disorders) | 1 (1)
Lightheadedness (General disorders) | 2 (2)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Damage to lead during procedure (e.g. accidental cut to lead body during pocket revision, device rep (Surgical and medical procedures) | 1 (1)
Hematoma (Surgical and medical procedures) | 3 (3)
Inability to successfully implant Protego lead due to patient anatomy (Surgical and medical procedures) | 1 (1)
Pocket pain (Surgical and medical procedures) | 1 (1)
RA lead dislodgement during a procedure (Surgical and medical procedures) | 1 (1)
RV lead dislodgement during a procedure (Surgical and medical procedures) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1)
Venous thrombosis without pulmonary embolism (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT02243696/Prot_SAP_000.pdf